CLINICAL TRIAL: NCT03884023
Title: Effect of REST on Cognitive Function and Hippocampus in the Alzheimer Disease Continuum
Brief Title: Effect of REST in the Alzheimer Disease Continuum
Acronym: ERADC
Status: Completed | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, Clinical Professor, Dongzhimen Hospital, Beijing
Other Study IDs: DZMEC-KY-2019-11
Record Dates: First submitted 2019-02-15; First posted 2019-03-21 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer's Disease
Keywords: Plasma REST; REST gene polymorphism; AD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AD group: Alzheimer's disease
- aMCI group: Amnestic Mild Cognitive(MCI) impairment due to Alzheimer's disease
- NC group: Normal Control

SUMMARY:
The investigators assume that REST gene polymorphism affects REST protein concentration, and REST protein concentration in peripheral blood is related to cognitive function and hippocampus. In this current study, REST protein content and gene polymorphism will be obtained in peripheral blood in AD and normal control. The effect of REST gene polymorphism on REST protein concentration will be discovered.The relationship between REST protein concentration and cognitive function will be found, as well as the relationship between REST protein concentration and hippocampus.

DETAILED DESCRIPTION:
Repressor element silencing transcription factor(REST), also known as neuron-restrictive silencer factor (NRSF) is a zinc finger protein of 121 kD and belongs to the Gli-Kruppel family with transcriptional regulation.This will be a Case-Crossover research. Consecutive participants will be divided into Alzheimer's disease dementia group, mild cognitive impairment due to Alzheimer's disease group and normal control group according to inclusion criteria of this research. Peripheral blood samples will be retained to detect REST gene polymorphisms and protein concentrations. Participants perform neuropsychological tests to assess cognitive function. Medial temporal atrophy scale is used to describe hippocampus. Differences in the mean or proportions between these 3 groups will be checked by t test or test. The relationship between REST protein concentration and cognitive function will be estimated, as well as the relationship between REST protein concentration and hippocampus.

ELIGIBILITY:
1. Inclusion Criteria of Normal Control (NC):

1. No active neurological and mental illness;
2. No use of psychotropic drugs;
3. Patients may have diseases, but these diseases and their treatment have no effect on cognition (MMSE>28);
4. Single cognitive field test was normal;
5. The clinical dementia rating scale is normal (CDR=0);
6. Aged 55-85, male or female;
7. Sufficient vision and hearing for neuropsychological tests;
8. Have a certain level of education, can read and write simple sentences;
9. Sign the informed consent.

2. Inclusion Criteria of AD-induced MCI (aMCI):

1. Complained of memory loss or/and confirmed by others;
2. Objective evidence suggests memory impairment (DSR<12.5 or HVLT<18.5, adjusted for age);
3. Preservation of overall cognitive function (MMSE 24-30/30, corrected according to education);
4. Most of daily life activities are reserved (ADL<16/56);
5. No dementia (CDR ≤0.5), and memory score was 0.5 or 1point;
6. Visual score of medial temporal atrophy (MTA) in MRI is greater than or equal to 0.5 or 1.0 point, which shall be corrected according to age);
7. Aged 55-85, male or female;
8. Sufficient vision and hearing for neuropsychological tests;
9. Sign the informed consent.

3. Exclusion Criteria of MCI due to AD:

1. Meet the DSM-IV diagnostic criteria of dementia;
2. Obvious cerebrovascular diseases in MRI;
3. Depression or other mental illnesses that meet the DSM-IV criteria in the past 2 years, the simplified version of the Geriatric Depression Scale (GDS-15) ≥ 8 ;
4. A history of alcohol or substance abuse or addiction in the past 2 years;
5. History of schizophrenia;
6. Any obvious neurological diseases, such as Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumors, progressive supra nuclear paralysis, epilepsy, chronic subdural hematoma, multiple sclerosis, severe head trauma with persistent neurological impairment or known structural brain abnormalities;
7. In investigator's impression, the subject cannot cooperate with the research procedure;
8. Other known systemic diseases that cause dementia (such as hypothyroidism, folate or vitamin B deficiency, neurosyphilis, HIV infection).

4. Inclusion Criteria for AD:

1. An insidious onset of disease in which symptoms develop gradually over months or years rather than suddenly over hours or days;
2. Definite history of cognitive deterioration was reported or observed;
3. Objective evidence suggests that at least one cognitive domain decline (e.g., DSR<9.5 or HVLT<18.5, adjusted for age);
4. Decrease in overall cognitive function (MMSE≤26, adjusted for education);
5. Decreased in ability of daily life: ADL≥16;
6. Dementia (CDR≥0.5), and memory score≥ 0.5;
7. Visual score of medial temporal atrophy in MRI (MTA) is greater than or equal to 0.5 or 1.0 point, adjusted for age);
8. Aged 55-85, male or female;
9. Sufficient vision and hearing for neuropsychological tests;
10. Sign the informed consent.

5. Exclusion Criteria for AD :

1. With severe cerebrovascular disease, defined as a history of stroke temporal associated with the occurrence or deterioration of cognitive impairment; Or the occurrence of multiple or severe infarction or severe white matter high signal;
2. Have the core characteristics of Lewy body dementia rather than dementia itself;
3. Significant characteristics of frontotemporal dementia with behavioral variation;
4. Significant characteristics of primary progressive semantic aphasia or primary progressive non-fluency/grammatical confusion aphasia;
5. Evidence of other complications of active neurological diseases, or non-neurological complications, or serious cognitive effects of drug use;
6. Depression or other mental illnesses that meet the DSM-IV criteria in the past 2 years, the simplified version of the Geriatric Depression Scale (GDS-15) ≥ 8 points;
7. Other known systemic diseases that cause dementia (such as hypothyroidism, folate or vitamin B deficiency, neurosyphilis, HIV infection).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population include Alzheimer's disease patients ,patients with amnestic mild cognitive impairment, and normal subjects who meet the inclusion and exclusion criteria and signed the informed consent in this study,and they will be recruited form outpatients, inpatients of Dongzhimen hospital and community.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of Gene polymorphism in rs2227902 and rs3796529. | baseline
  Verifying the value of REST gene polymorphism as an early markers of Alzheimer's Disease
Concentration of REST protein | baseline
  Verifying the value of REST protein detection as an early markers of Alzheimer's Disease

CONTACTS AND LOCATIONS:
Overall Officials: Tian Jinzhou, MD,PhD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China